CLINICAL TRIAL: NCT00689624
Title: A Triplet Combination With Irinotecan Plus Oxaliplatin,Continuous Infusion 5-Fluorouracil And Leucovorin Plus Cetuximab As First Line Treatment In Metastatic Colorectal Cancer. A Pilot Phase II Trial
Brief Title: Irinotecan/Oxaliplatin/5-Fluorouracil/Leucovorin/Cetuximab As First Line Treatment In Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, MD, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.21
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Cetuximab; FOLFOXIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Leucovorin; Oxaliplatin; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): FOLFOXIRI+Erbitux
  Interventions: Drug: Irinotecan; Drug: Leukovorin; Drug: Oxaliplatin; Drug: 5-FLUOROURACIL; Drug: Cetuximab

INTERVENTIONS:
Drug: Irinotecan — Irinotecan will be administered at a dose of 150mg/m2 as a 30 min IV infusion on day 1
  Other Names: CPT-11; Campto
Drug: Leukovorin — Leukovorin will be administered at a dose of 200mg/m2 as a 2-hour IV infusion on days 2 and 3
  Other Names: LV
Drug: Oxaliplatin — Oxaliplatin will be administered on day 2 at the dose of 65mg/m2 as a 2-hours IV
  Other Names: LoHP; Eloxatin
Drug: 5-FLUOROURACIL — 5-FLUOROURACIL at the dose of 400mg/m2 as IV bolus and then, 600mg/m2 as a 22-hour continuous IV infusion, on days 2 and 3
  Other Names: 5-FU
Drug: Cetuximab — Cetuximab will be administered at the dose of 500mg/m2 as a 2-hour infusion on day 1 at least one hour before chemotherapy
  Other Names: Erbitux

SUMMARY:
This study will evaluate the efficacy of FOLOFOXIRI plus Cetuximab combination in young patients with good performance status with unresectable metastatic colorectal cancer.

DETAILED DESCRIPTION:
The combination of FOLFOXIRI plus cetuximab is reasonable safe regimen especially for patients with good performance status. The estimated benefit from the combination is greater than the possible risk, especially for the patients who will become resectable after treatment. It will be extremely interesting to evaluate the resectability rate of this specific group of patient with good performance status and unresectable disease when they are treated with all active chemotherapeutic agents and cetuximab

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven metastatic adenocarcinoma of the colon or rectum
* Previous chemotherapy for metastatic disease not allowed. Patients who received prior adjuvant 5-FU-based chemotherapy are eligible if they have remained free of disease for at least 6 months after the completion of adjuvant therapy
* Patients with operable metastatic disease are excluded from the study
* Age 18-70 years
* Performance status (ECOG) 0-1
* At least one bidimensionally measurable lesion of >= 2cm
* Life expectancy of at least 6 months
* Adequate hematologic parameters (absolute neutrophil count >= 1.5x109/L and platelets >=100x109/L)
* Creatinine and total bilirubin < 1.25 times the upper limit of normal
* Aspartate and alanine aminotransferase < 3.0 times the upper limit of normal (<5 times in case of liver mets)

Exclusion Criteria:

* Absence of active infection or malnutrition (loss of more than 20% of the body weight)
* No history of a second primary tumor other than non-melanoma skin cancer or in situ cervical carcinoma. curatively treated
* Patients treated with palliative radiotherapy had to have measurable metastatic disease outside the irradiation fields.
* Patients with severe cardiac dysfunction, liver metastases involving more than 50% of the liver parenchyma, chronic diarrhea, or prior irradiation affecting more than 30% of the active bone marrow are excluded.
* All patients will have to sign written informed consent in order to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 2 months

SECONDARY OUTCOMES:
Resectability rates | Resectability at the end of treatment (4 or 6 months from the entry to the study)
Time to Tumor Progression | 1 year
Overall Survival | 1 year
Toxicity profile | Toxicity assessment on each chemotherapy cycles (every 15 days)
Pharmacogenomic analysis | During the treatment
Q-Twist analysis of Quality of life | Quality of life assessment every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Crete
Locations (1):
- University Hospital of Crete, Heraklion, Greece